CLINICAL TRIAL: NCT06612463
Title: Effect of Caffeine Supplementation on Movement Patterns and Reactive Agility in Rugby Sevens Matches
Brief Title: Caffeine Supplementation on Movement Patterns and Reactive Agility in Rugby Sevens Matches
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chen Kang, Professor, National Taiwan Sport University
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 111-03; MOST 111-2410-H-028-002-MY3 (Other Grant/Funding Number: National Science and Technology Council, Taiwan)
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Exercise
Keywords: caffeine; rugby sevens; global positioning system
MeSH Terms: conditions — Motor Activity | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: 2 types of Intervention: caffeine or placebo. Arm 1: Caffeine trial: Participants ingested a capsule containing 3 mg/kg caffeine (Wako Pure Chemical Industries, Ltd., Osaka, Japan) 60 min prior to the match.
  Arm 2: Placebo trial: Participants ingested a capsule containing starch (Chung-Yu Biotech Co LTD, Taichung, Taiwan) at the same time point.
  The capsules used in both trials were identical in appearance. The caffeine and placebo supplements were prepared by a laboratory technician who was independent of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The capsules used in both trials were identical in appearance. The caffeine and placebo supplements were prepared by a laboratory technician who was independent of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): In the caffeine trial, participants ingested a capsule containing 3 mg/kg caffeine (Wako Pure Chemical Industries, Ltd., Osaka, Japan) 60 min prior to the match.
  Interventions: Dietary Supplement: Caffeine 6mg/kg
- Placebo (Placebo Comparator): In the placebo trial, participants ingested a capsule containing starch (Chung-Yu Biotech Co LTD, Taichung, Taiwan) at the same time point.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine 6mg/kg — In the caffeine trial, participants ingested a capsule containing 3 mg/kg caffeine 60 min prior to each rugby sevens match. There was 2 matches per day. So the total dosage is 6 mg/kg/ day
  Arms: Caffeine
Dietary Supplement: Placebo — In the placebo trial, participants ingested a capsule containing starch 60 min before each rugby sevens match. There were 2 matches per day
  Arms: Placebo

SUMMARY:
Caffeine is widely used by rugby players for its performance-enhancing effects. The main questions it aims to answer are: (1) the impact of caffeine supplementation on various performance metrics, including distance covered at different speeds, acceleration, deceleration, collisions, and repeated high-intensity efforts; and (2) reactive agility, across four matches over two consecutive days in collegiate male rugby sevens players.A position-matched, double-blind, randomized crossover design was employed, with six male collegiate rugby players (mean height: 1.78 ± 0.09 m, mean weight: 81.3 ± 9.2 kg) participating in two trials. Each trial consisted of a two-day tournament, with two matches per day. Movement was monitored using global positioning system units.

DETAILED DESCRIPTION:
This study employed a position-matched, double-blind, randomized crossover design. Pairs of participants with similar playing positions, specifically forwards or backs/scrum halves, were randomly assigned to either the caffeine or placebo trial. Each trial comprised a two-day rugby sevens tournament, with participants playing two matches per day. Following a 13-day washout period, participants switched to the alternate trial. Both the participants and the research personnel were blinded to the supplementation condition throughout the study period, with the assignment of supplements disclosed to research personnel only after all data analyses were completed.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone regular rugby training for at least three years
* Member of a Division I university rugby team

Exclusion Criteria:

* Musculoskeletal injury within one month prior to the study
* Presence of major cardiovascular diseases
* Presence of major metabolic diseases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Total Distance and Distance Covered in Speed Zones | Each trial contained 2 days, with 2 matches on each day. Each participant completed 2 trials
  This variable was measured with wearable global positioning system device during rugby sevens matches. Speed is divided into six zones: standing and walking (0-6 km/h), jogging (6-12 km/h), cruising (12-14 km/h), striding (14-18 km/h), high-intensity running (18-20 km/h), and sprinting (> 20 km/h). The distance covered in each speed zone and the total distance covered were recorded.
Acceleration and Deceleration | Each trial contained 2 days, with 2 matches on each day. Each participant completed 2 trials
  This variable was measured with wearable global positioning system device during rugby sevens matches. For an activity to be included in the analysis, the movement speed must exceed 5 km/h, and the acceleration must be greater than 2 m/s² or the deceleration must be less than -2 m/s², sustained for more than 0.9 s. If the interval between two movements is less than 1 s, the subsequent movement will be combined with the previous one for analysis. The frequency and distance covered during these acceleration and deceleration phases were recorded.
collision | Each trial contained 2 days, with 2 matches on each day. Each participant completed 2 trials
  This variable was measured with wearable global positioning system device during rugby sevens matches. Collision is defined as the number of times a participant accumulates 0.5 s standing after body contact resulting in a fall. Specific collision events include rucks, tackles, and instances where a player falls after contact
Repeated High-Intensity Effort | Each trial contained 2 days, with 2 matches on each day. Each participant completed 2 trials
  This variable was measured with wearable global positioning system device during rugby sevens matches. A repeated high-intensity effort is defined as the completion of three or more high-intensity actions in succession, with rest periods of no more than 21 s between each action. The criteria for high-intensity actions include a movement speed of at least 14 km/h, an acceleration of at least 2 m/s², and a deceleration of at least -2 m/s²
Reactive Agility | Each trial contained 2 days, with 2 matches on each day. Reactive agility was measured before each match. Each participant completed 2 trials
  The participants sprinted with the ball, passing through a light gate, after which an indicator light immediately displayed a left or right direction. The participants had to respond by changing direction according to the indicator and continue moving until they passed the second light gate positioned 1.5 m away from the indicator. The fastest time from two attempts was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kang Chang, PhD, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Del Coso J, Portillo J, Munoz G, Abian-Vicen J, Gonzalez-Millan C, Munoz-Guerra J. Caffeine-containing energy drink improves sprint performance during an international rugby sevens competition. Amino Acids. 2013 Jun;44(6):1511-9. doi: 10.1007/s00726-013-1473-5. Epub 2013 Mar 5. PMID 23462927